CLINICAL TRIAL: NCT02892695
Title: PCAR-119 Bridge Immunotherapy Prior to Stem Cell Transplant in Treating Patients With CD19 Positive Relapsed or Refractory Leukemia and Lymphoma
Brief Title: PCAR-119 Bridge Immunotherapy Prior to Stem Cell Transplant in Treating Patients With CD19 Positive Leukemia and Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Hefei (Other); Hefei Binhu Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-119-001
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Follicular Lymphoma; Mantle Cell Lymphoma; B-cell Prolymphocytic Leukemia; Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Prolymphocytic, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Sensitivity and Specificity; Antigens, CD19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR-NK Cell immunotherapy (Experimental): Enrolled patients will receive CAR-NK cell immunotherapy with a novel specific chimeric antigen receptor targeting CD19 antigen by infusion.
  Interventions: Biological: anti-CD19 CAR-NK cells

INTERVENTIONS:
Biological: anti-CD19 CAR-NK cells — The allogeneic NK cells (NK-92 cell line for clinical use) are engineered to contain anti-CD19 attached to TCRzeta, CD28 and 4-1BB signaling domains. These modified cells are called chimeric antigen receptor NK cells with specificity for CD19.
  Other Names: chimeric antigen receptor NK cells with specificity for CD19

SUMMARY:
The purpose of this study is to evaluate the safety and optimal dose of PCAR-119 in patients who are going to receive stem cell transplantation but without available treatment to achieve complete remission prior to the transplant.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and optimal dose of PCAR-119 in patients who are going to receive stem cell transplantation but without available treatment to achieve complete remission prior to the transplant. In addition, some patients who enroll to other CD19-CAR-T cell therapy trials might be eligible for this trial if their CD19-CAR-T cells cannot be produced successfully because they have insufficient T cells to allow the CD19-CAR-T cells to be made; their T cells are inefficiently transduced with CAR viruses; or their CAR-T cell expansion is failed.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects with CD19+ B cell malignancies in patients who have no available curative treatment options except stem cell transplantation, with limited prognosis (several months to < 2 year survival) and no available treatment option to achieve complete remission prior to transplant. Some patients who have enrolled to other CD19-CAR-T cell therapy trials may be eligible if their CD19-CAR-T cells cannot be produced successfully because they have insufficient T cells to allow the CD19-CAR-T cells to be made; their T cells are inefficiently transduced with CAR viruses; or their CAR-T cell expansion is failed. All of those patients must meet the following criteria:

1. Eligible diseases: Acute lymphocytic leukemia (ALL), Chronic lymphocytic leukemia (CLL), Follicular lymphoma, Mantle cell lymphoma, B-cell prolymphocytic leukemia, and diffuse large cell lymphoma, previously identified as CD19+.
2. Patients 3 years of age or older, and must have a life expectancy > 12 weeks.
3. Eastern cooperative oncology group (ECOG) performance status of 0-2 or karnofsky performance status (KPS) score is higher than 60.
4. Females of child-bearing potential must have a negative pregnancy test and all subjects must agree to use an effective method of contraception for up to two weeks after the last infusion of CAR NK cells.
5. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: White blood cell count (WBC) ≥ 2500c/ml, Platelets ≥ 50×10^9/L, Hb ≥ 9.0g/dL, lymphocyte (LY) ≥ 0.7×10^9/L, LY% ≥ 15%, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5×upper limit of normal, serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration.
6. Ability to give informed consent.

Exclusion Criteria:

1. Pregnant or nursing women may not participate.
2. Active HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at the time of screening.
3. Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.
4. History of severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, or aldesleukin.
5. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
6. The existence of unstable or active ulcers or gastrointestinal bleeding.
7. Patients need anticoagulant therapy (such as warfarin or heparin).
8. Patients need long-term antiplatelet therapy (aspirin at a dose > 300mg/d; clopidogrel at a dose > 75mg/d).
9. Patients using fludarabine or cladribine chemotherapy within 3 months prior to leukapheresis.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events attributed to the administration of the anti-CD19 CAR-NK cells | 2 years

SECONDARY OUTCOMES:
Objective Response Rate | Safety follow-up is 100 days from last CAR-NK infusion

CONTACTS AND LOCATIONS:
Locations (1):
- PersonGen BioTherapeutics (Suzhou) Co., Ltd., Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Del Zotto G, Marcenaro E, Vacca P, Sivori S, Pende D, Della Chiesa M, Moretta F, Ingegnere T, Mingari MC, Moretta A, Moretta L. Markers and function of human NK cells in normal and pathological conditions. Cytometry B Clin Cytom. 2017 Mar;92(2):100-114. doi: 10.1002/cyto.b.21508. Epub 2017 Feb 12. PMID 28054442